CLINICAL TRIAL: NCT04058197
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study of the Safety and Efficacy of Deferoxamine Intradermal Delivery Patch (DIDP) in Chronic Sickle Cell Leg Ulcers
Brief Title: Deferoxamine for Sickle Cell Chronic Leg Ulcer Treatment
Acronym: D-SCOUT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: TauTona Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CD1001
Record Dates: First submitted 2019-06-18; First posted 2019-08-15 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2020-11

CONDITIONS: Chronic Cutaneous Ulcer; Sickle Cell Disease
Keywords: chronic sickle cell leg ulcer
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Deferoxamine (DFO) Intradermal Delivery Patch (DIDP), 45mg DFO daily, up to 12 weeks
  Interventions: Drug: Deferoxamine Product
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Deferoxamine Product — Deferoxamine Intradermal Delivery Patch
  Arms: Active
Other: Placebo — Placebo Patch
  Arms: Placebo

SUMMARY:
Approximately 60 subjects will be enrolled into this double-blind, placebo-controlled study for the Deferoxamine Intradermal Delivery Patch (DIDP).

Those subjects who pass Screening will enter into the 2-week Standard of Care (SOC) Run-In period. During this time, ulcers will be assessed to check healing based on digital planimetry, and qualitative features of the ulcer. Subjects who meet eligibility criteria at the end of the 2-week Run-in Period will be randomized into active and control groups (2 active to 1 placebo) and enter the 12-week Treatment Period. At each visit during the Treatment Period, the target ulcer will be measured by digital photographic planimetry, the Principal Investigator will assess the wound qualitative attributes, and the DIDP (or placebo patch) will be placed as the primary wound dressing. At each visit the subject will also receive/review a daily diary to document pain , study drug compliance, and analgesic use.

DETAILED DESCRIPTION:
Approximately 60 subjects will be enrolled to allow for up to 48 male or female subjects with SCD and cutaneous ulcers to complete this double-blind, placebo-controlled study.

A sentinel group of 3 subjects will be enrolled and evaluated for safety (while still blinded). The remaining subjects will be enrolled in a 2:1 ratio, active:placebo.

Those subjects who pass Screening will enter into the Standard of Care (SOC) Run-In period. During this time, ulcers will be assessed to check healing based on digital planimetry, and qualitative features of the ulcer. Subjects who meet eligibility criteria at the end of the Run-in Period will be randomized and enter the 12-week Treatment Period.

The DIDP (or placebo) will be replaced daily at home. The subject will visit the clinic on an approximately weekly basis for study assessments, to include imaging and planimetric wound measurements and qualitative wound assessments. Clinical laboratory samples will be collected at Treatment Baseline, Treatment Weeks 4, 8 and 12, or at End of Study (EOS) visit if sooner. A blood sample for PK testing will also be collected at these timepoints. During this Treatment Period, if at any time the wound has met the criterion for 100% healing, the subject will immediately go into the 4-week Follow-up Period.

During the Follow-up Period, the subject will come to the clinic at 1-week intervals. At these visits, the area of the wound will continue to be protected with a protective dressing. Clinical laboratory samples will be collected at the Termination Visit.

Ulcer pain will be assessed by the subject daily and recorded in a diary, along with a record of analgesic use. At each visit, study staff will assist the subjects to assign an overall ulcer pain score for the week.

Quality of Life Assessment will be performed at Baseline prior to dosing and at End of Treatment.

Safety will be assessed based upon known adverse outcomes of Deferoxamine (DFO) therapy. Skin will be examined for evidence of rash and skin irritation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >18 years of age
2. Diagnosed with Sickle Cell Disease (SS, SC, Sß-thalassemia, SD, SOArab)
3. Cutaneous ulcer with a University of Texas Wound Classification System Grade 1A or 2A (= Wagner class 1or 2, without infection or ischemia)
4. Ulcer on lower leg, ankle, or dorsum of foot
5. Vascular status of site assessed and judged adequate for healing (per Section 4.2)
6. Ulcer present ≥ 14 days but not > 6 months at time of screening
7. Ulcer 2.0 cm2 to 45.0 cm2 and < 6.0 cm diameter at widest point after debridement, prior to randomization.
8. Ulcer healed by < 25% during the SOC run-in period prior to Visit 4 randomization.
9. Subject is willing to use acceptable form of birth control (per Section 4.2) during trial and for one month thereafter

Exclusion Criteria:

1. Active infection/purulence at ulcer site, based on Investigator's clinical judgement
2. Current or history of osteomyelitis at or near site of ulcer
3. Serum albumin < 2.0 g/dL
4. Treatment with systemic DFO within 7 days of study entry
5. Serum ferritin > 1000 ng/mL
6. Subjects requiring, or expected to require, iron chelation therapy (systemic deferoxamine, deferasirox, or deferiprone) during the duration of the study.
7. Subjects on dialysis or with evidence of nephrotic syndrome.
8. Known bleeding or coagulation disorder that would preclude surgical debridement, as necessary.
9. The subject has a major uncontrolled medical disorder, such as serious cardiovascular, renal, liver, pulmonary disease, or pulmonary disease (per Investigator discretion).
10. Any condition that in the Investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study
11. Previous participation in another clinical trial within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety / Tolerability] | 12 weeks
  Incidence of systemic and local adverse events of DIDP applied to non-healing cutaneous leg ulcers. Changes from baseline characteristics that are treatment-related as measured by physical examinations, clinical laboratory, skin and other physiologic assessments.

SECONDARY OUTCOMES:
Degree of Wound closure | 12 weeks
  Percentage of wound closure
Partial wound closure incidence | 12 weeks
  Incidence of 80% closure
Total wound closure incidence | 12 weeks
  Incidence of 100% closure
Wound closure rate | 12 weeks
  rate of closure
Ulcer recurrence | 4 week follow-up post
  Incidence

OTHER OUTCOMES:
Ulcer pain: Numeric Pain Rating Scale | 12 weeks
  Numeric Pain Rating Scale (McCaffery et al, 1989) Scale: 0-10 (0 = no pain, 10 = severe pain)
Analgesic use | 12 weeks
  Diary: Opioid analgesic use converted as morphine mg equivalents (MME). Non-steroidal use will be descriptive.
QOL: Health-related QOL in Chronic Wounds | 12 weeks
  Wound QOL: Health-related QOL in Chronic Wounds (Augustin et el, 2014; Blome et al, 2014) Response range: "not at all" -to- "very much"
Pharmacokinetics (blood) | 12 weeks
  Deferoxamine / Placebo Peak plasma concentration (Cmax)
Pharmacokinetics (blood) | 12 weeks
  Deferoxamine / Placebo Time of peak plasma concentration (Tmax)
Pharmacokinetics (blood) | 8 hours
  Deferoxamine / Placebo Plasma concentration over 8 hours

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Miami, Miami, Florida
  - Sonar Clinical Research LLC, Atlanta, Georgia
  - Montefiore Medical Center, The Bronx, New York